CLINICAL TRIAL: NCT02182700
Title: Open Study on the Efficacy and Safety of Combivent® Aerosol (120 mcg Salbutamol Sulfate Plus 20 mcg Ipratropium Bromide) + Spacer, 12 to 24 Puffs, in Adult Patients With Moderate to Severe Asthma Crisis
Brief Title: Efficacy and Safety of Combivent® Aerosol and Spacer, in Adult Patients With Moderate to Severe Asthma Crisis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1012.32
Record Dates: First submitted 2014-07-03; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol; Ipratropium

ARMS (1):
- Combivent® aerosol (Experimental)
  Interventions: Drug: salbutamol sulfate + ipratropium bromide

INTERVENTIONS:
Drug: salbutamol sulfate + ipratropium bromide — 120 mcg (salbutamol sulfate) + 20 mcg (ipratropium bromide), inhalation (metered aerosol plus spacer)
  Other Names: Combivent® aerosol

SUMMARY:
Study to evaluate the bronchodilator efficacy and safety of a fixed combination of salbutamol sulfate (120 mcg) + ipratropium bromide (20mcg) (Combivent® MDI) in aerosol plus spacer in adult patients with moderate-to-severe asthma crisis who arrived at the emergency room.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with a diagnosis of asthma according to the American Thoracic Society (ATS) presenting at the emergency room with an acute moderate and/or severe asthma attack
* Patients aged between18 to 40 years
* Patients able to perform spirometry (PEFR and FEV1)
* PEFR < 60% and > 25 % of predicted normal value or a FEV1 <= 60% of predicted normal value
* Patients able to sign witnessed informed consent

Exclusion Criteria:

* Patients with very severe or life threatening obstruction, manifested by:

  * Cyanosis of tongue and lips
  * Confusion, drowsiness, coma or exhaustion
  * Silent chest on auscultation or weak respiratory effort
  * PEFR < 25% the predicted normal value
  * Bradycardia (of less 60 beats/min)
* Patients with a smoking history of more than 10 pack/years
* Patients with chronic obstructive pulmonary disease (COPD)
* Patients on treatment for or suspected as having glaucoma
* Patients with uncontrolled hypertension
* Patients with known allergy or contra-indications to either salbutamol, ipratropium or hydrocortisone or their excipients
* Female patients known or suspected to be pregnant or nursing
* Patients known or suspected on clinical grounds to have pneumonia, pneumothorax or pneumomediastinum
* Patients with a history of chest surgery
* Patients with other respiratory conditions if diagnosed. These included pulmonary fibrosis, bronchiectasis, cystic fibrosis, pulmonary tuberculosis, pulmonary complications of AIDS, lung cancer
* Patients requiring drugs for the treatment of the acute asthma attack other than the study drug, hydrocortisone or oxygen
* Patients who have previously recruited into this study
* Patients who have been on other investigational drugs within three months prior to study entry
* Patients with acute myocardial infarction, pulmonary edema or other life threatening disease, which in the judgment of the ER (Emergency room) physician precluded entry into the study
* Patients with obvious or previous diagnosed serious hepatic or renal impairment or bladder neck obstruction

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 1998-07; Primary Completion 1999-12 (Actual)

PRIMARY OUTCOMES:
Number of patients discharged with a peak flow expiratory flow rate (PEFR) >= 70% predicted normal value at the end of the first and the second treatment | 60 and 120 min after starting treatment

SECONDARY OUTCOMES:
Number of patients whose PEFR >= 60% within the first or the second hour | 60 and 120 min after start of treatment
Hospitalisation period at the Intensive Care Unit (ICU) | up to 3rd hour after treatment
Hospitalisation time at the general ward | up to 3rd hour after treatment
Number of relapses and/or new episodes | 7 days after finishing treatment